CLINICAL TRIAL: NCT04108156
Title: A Phase III, Multicenter, Randomized, Visual Assessor-Masked, Active-comparator Study of the Efficacy, Safety, and Pharmacokinetics of the Port Delivery System With Ranibizumab in Patients With Diabetic Macular Edema (Pagoda)
Brief Title: A Study to Evaluate Efficacy, Safety & Pharmacokinetics of the Port Delivery System (PDS) With Ranibizumab in Participants With Diabetic Macular Edema (DME) Compared With Intravitreal Ranibizumab; A Substudy to Evaluate the Safety of Re-implanting the PDS With Ranibizumab in Participants With DME
Acronym: Pagoda
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GR40550
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Diabetic Macular Edema
Keywords: Port Delivery System
MeSH Terms: interventions — Ranibizumab; Injections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The substudy is a non-randomized, open-label study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- PDS Arm (Experimental): Participants randomized to the PDS arm will receive IVT ranibizumab injection Q4W (loading phase) and will then have the PDS implant (pre-filled with ranibizumab) surgically inserted. PDS implant refill-exchange procedures will be performed on a fixed interval Q24W thereafter.
  Interventions: Drug: PDS Implant Pre-Filled with 100 mg/mL Ranibizumab; Drug: Ranibizumab refill exchange
- Intravitreal Arm (Active Comparator): Participants randomized to the intravitreal arm will receive IVT ranibizumab injection Q4W until they receive the PDS implant (pre-filled with ranibizumab). PDS implant refill-exchange procedures will be performed on a fixed interval Q24W thereafter.
  Interventions: Drug: Intravitreal Ranibizumab 0.5 mg Injection; Drug: Ranibizumab refill exchange
- Substudy: Cohort 1 (Experimental): Participants will undergo re-implantation with the updated PDS implant (pre-filled with ranibizumab 100 milligrams per milliliter [mg/mL]) on Day 1 (or enrollment visit) and then will have two refill-exchanges (ranibizumab 100 mg/mL) Q24W up to 48 weeks.
  Interventions: Drug: PDS Implant Pre-Filled with 100 mg/mL Ranibizumab; Drug: Ranibizumab refill exchange
- Substudy: Cohort 2a (Experimental): Participants who received an updated PDS implant, have < 24 weeks post-re-implantation follow-up and no scheduled refill-exchange visit in the main study, will undergo two refill-exchange procedures (ranibizumab 100 mg/mL) Q24W, post main study re-implantation visit.
  Interventions: Drug: Ranibizumab refill exchange
- Substudy: Cohort 2b (Experimental): Participants who received an updated PDS implant, have < 48 weeks post-re-implantation follow-up and one refill exchange visit in the main study, regardless of whether the refill exchange was administered or the visit was missed, will undergo one refill-exchange procedure (ranibizumab 100 mg/mL) Q24W, post main study re-implantation visit.
  Interventions: Drug: Ranibizumab refill exchange

INTERVENTIONS:
Drug: PDS Implant Pre-Filled with 100 mg/mL Ranibizumab — Will be administered as per the schedule described in individual arm.
  Arms: PDS Arm; Substudy: Cohort 1
Drug: Intravitreal Ranibizumab 0.5 mg Injection — Will be administered as per the schedule described in individual arm.
  Arms: Intravitreal Arm
Drug: Ranibizumab refill exchange — Will be administered as per the schedule described in individual arm.

SUMMARY:
This study will evaluate the efficacy, safety, and Pharmacokinetics (PK) of the PDS with ranibizumab in participants with DME when treated every 24 weeks (Q24W) compared with intravitreal (IVT) ranibizumab 0.5 milligrams (mg) every 4 weeks (Q4W).

The substudy will evaluate safety of re-implanting the updated PDS with ranibizumab and the refill-exchange procedures following re-implantation in participants with DME who were previously enrolled in the main study, GR40550. Up to 100 participants from the main study will be enrolled and followed for a maximum of 72 weeks post-re-implantation in the substudy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at time of signing informed consent form (ICF)
* Documented diagnosis of diabetes mellitus (Type 1 or Type 2)
* Glycated haemoglobin (HbA1c) level of ≤10% within 2 months prior to screening or at screening

Study eye

* Macular thickening secondary to DME involving the center of the fovea with CST ≥325 micrometer (µm) on SD-OCT at screening
* BCVA score of 78 to 25 letters (20/32 to 20/320 approximate Snellen equivalent)

Exclusion Criteria:

* High-risk PDR
* Active intraocular inflammation (grade trace or above)
* Suspected or active ocular or periocular infection of either eye
* Uncontrolled ocular hypertension or glaucoma and any such condition the investigator determines may require a glaucoma-filtering surgery during a patient's participation in the study
* Cerebrovascular accident or myocardial infarction within 6 months prior to randomization
* Atrial fibrillation diagnosis or worsening within 6 months prior to randomization
* Uncontrolled blood pressure

Substudy:

Inclusion Criteria:

* Having experienced a septum dislodgement in the original implant while in the main study or after exiting the main study
* Sufficiently clear ocular media and adequate pupillary dilation to allow for analysis and grading by central reading center

Exclusion Criteria (Cohort 1 Only):

* Recent history (in the last 3 months prior to enrollment) of other disease, other non-diabetic metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a condition that contraindicates the use of ranibizumab or surgical placement of the PDS implant; that might affect interpretation of the results of the study; or that renders the participant at high risk for treatment complications
* Active cancer within the last 12 months, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or prostate cancer
* Current systemic treatment for a confirmed active systemic infection
* Participation in an investigational trial that involves treatment with any drug or device (with the exception of vitamins and minerals or enrollment in Study GR40550) within 6 months prior to enrollment
* Use of antimitotic or antimetabolite therapy within 30 days

Ocular Exclusion Criteria for Study Eye:

* Any ocular condition that may render the participant at high risk for surgical or treatment complications
* Intraocular surgery (including cataract surgery) within 1 month preceding the enrollment visit
* Any use of medicated intraocular implants (other than the PDS implant), at any time prior to enrollment
* History of rhegmatogenous retinal tears or peripheral retinal breaks within 3 months prior to the enrollment visit
* Any concurrent ocular condition that would require surgical intervention during the study to prevent or treat visual loss
* Concurrent conjunctival, tenon's capsule, and/or scleral condition in the supero-temporal quadrant of the eye (e.g., scarring, thinning, mass) that may affect the refill-exchange procedure of the PDS implant
* Ongoing ocular complications that might affect participant safety Ocular Exclusion Criteria for Either Eye
* Suspected or active ocular or periocular infection (e.g., infectious conjunctivitis or endophthalmitis)
* Any history of uveitis
* Active blepharitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 634 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2027-11-16 (Estimated); Study Completion 2027-11-16 (Estimated)

PRIMARY OUTCOMES:
Change in BCVA Score From Baseline Averaged Over Weeks 60 and 64 as Measured Using the ETDRS Chart in the Efficacy Population Using a Treatment Policy Strategy for all Intercurrent Events | Baseline to Week 64
  BCVA = Best-Corrected Visual Acuity
  ETDRS = Early Treatment Diabetic Retinopathy Study
  A vision score of 20/20 vision is considered normal. A score of 20/200 is considered being legally blind.
Substudy: Number of Participants With Ocular and Systemic (Non-ocular) Adverse Events (AEs) and Severity of Ocular and Systemic AEs | Baseline to Week 72
Substudy: Number of Participants With Adverse Events of Special Interests (AESIs) and Severity of AESIs | Baseline to Week 72
Substudy: Duration of AESIs | Baseline to Week 72
Substudy: Number of Participants With Ocular AESIs and Severity of Ocular AESIs During the Post-operative Period | Up to Day 37 post re-implantation
Substudy: Number of Participants With Ocular AESIs and Severity of Ocular AESIs During the Follow-up Period | > 37 days post-implantation (up to approximately 72 weeks)
Substudy: Duration of Ocular AESIs During the Post-operative Period | Up to Day 37 post re-implantation
Substudy: Duration of Ocular AESIs During the Follow-up Period | > 37 days post-implantation (up to approximately 72 weeks)
Substudy: Number of Participants With Adverse Device Effects (ADEs) and Severity of ADEs | Baseline to Week 72
Substudy: Number of Participants With Anticipated Serious ADEs | Baseline to Week 72
Substudy: Duration of Serious ADEs | Baseline to Week 72
Substudy: Number of Device Deficiencies | Baseline to Week 72

SECONDARY OUTCOMES:
Change in BCVA Score From Baseline Averaged Over Weeks 60 and 64 as Measured With Use of the ETDRS Chart in the Modified Intent-to-treat (mITT) Population Using a Treatment Policy Strategy for All Intercurrent Events | Baseline to Week 64
  ETDRS-DRSS = ETDRS Diabetic Retinopathy Severity Scale
Change in BCVA Score From Baseline Averaged Over Weeks 60 and 64 as Measured With Use of the ETDRS Chart in the mITT Population Using a Hypothetical Strategy for All Intercurrent Events | Baseline to Week 64
Percentage of Participants With a ≥2-step Improvement From Baseline on the ETDRS-DRSS at Week 64 in the Efficacy Population | Baseline to Week 64
Percentage of Participants With a ≥2-step Improvement From Baseline on the ETDRS-DRSS at Week 64 in the mITT population | Baseline to Week 64
Change from Baseline in BCVA as Measured on the ETDRS Chart Over Time | Baseline up to Week 120
Percentage of Participants Who Lose <15, <10, and <5 letters in BCVA From Baseline Over Time | Baseline up to Week 120
Percentage of Participants Who Gain ≥15, ≥10, ≥5, ≥0 Letters in BCVA From Baseline Over Time | Baseline up to Week 120
Percentage of Participants With a BCVA Snellen Equivalent of 20/40 or Better Over Time | Baseline up to Week 120
Percentage of Participants With a BCVA Snellen Equivalent of 20/200 or Worse Over Time | Baseline up to Week 120
Percentage of Participants With a ≥2-step Improvement From Baseline on the ETDRS-DRSS Over Time | Baseline up to Week 120
Percentage of Participants With a ≥3-step Improvement From Baseline on the ETDRS-DRSS Over Time | Baseline up to Week 120
Time to ≥2-step Worsening From Baseline on the ETDRS-DRSS | Baseline up to Week 120
Time to ≥3-step Worsening From Baseline on the ETDRS-DRSS | Baseline up to Week 120
Change From Baseline in ETDRS-DRSS Score Over Time | Baseline up to Week 120
Change From Baseline in Central Subfield Thickness (CST) as Measured on Spectral Domain Optical Coherence Tomography (SD-OCT) Over Time | Baseline up to Week 120
Change From Baseline in Total Macular Volume as Measured on SD-OCT Over Time | Baseline up to Week 120
Percentage of Participants With Absence of Intraretinal Fluid (IRF) Over Time (IRF as Measured in the Central 1 mm Subfield) | Baseline up to Week 120
Percentage of Participants With Absence of Subretinal Fluid (SRF) Over Time (SRF as Measured in the Central 1 mm Subfield) | Baseline up to Week 120
Percentage of Participants With Absence of IRF and SRF Over Time | Baseline up to Week 120
Percentage of Participants With Absence DME (Defined as CST ≥325 μm on SD-OCT) Over Time | Baseline up to Week 120
  DME = diabetic macular edema
Time to PDR (Defined as a Score ≥60 on the ETDRS-DRSS) | Baseline up to Week 120
  PDR = proliferative diabetic retinopathy
Percentage of Participants Who do not Undergo Supplemental Treatment With IVT Ranibizumab Within Each Refill-exchange Interval | Baseline up to Week 120
Percentage of Participants Who Report Preferring PDS Treatment Compared With IVT Ranibizumab Treatment | Baseline to Week 64
  As measured by the PDS patient preference questionnaire (PPPQ) at Week 64 among participants in the PDS arm efficacy population, mITT population
Percentage of Participants Who Report Preferring PDS Treatment Compared With IVT Ranibizumab Treatment, as Measured by the PPPQ at Week 64 | Baseline to Week 64
  Participants in a subset of patients with bilateral disease who are simultaneously receiving ranibizumab via study eye PDS implant and fellow eye IVT injection.
Participant-reported Vision-related Functioning and Health-Related Quality of Life (HRQoL) Among Participants in Both Treatment Arms, as Measured by Changes From Baseline | , Baseline Week 48, Week 96
  As measured by in the National Eye Institute Visual Function Questionnaire-25 (NEI VFQ-25) composite score and Near Activities, Distance Activities, and Driving subscale scores
Participant-reported Vision-related Functioning and HRQoL, as Measured by the Proportion of Participants With a ≥ 4-Point Improvement From Baseline in the NEI VFQ-25 Composite Score at Weeks 48 and 96 Among Participants in Both Treatment Arms | Baseline, Week 48, Week 96
Incidence and Severity of Ocular AEs | Baseline to Week 120
Incidence and Severity of Non-ocular AEs | Baseline up to Week 120
Incidence, Severity, and Duration of AEs of Special Interest | Baseline up to Week 120
Serum Concentration of Ranibizumab Observed Over Time | Baseline up to Week 120
PK Parameter: Value Area Under the Concentration- Time Curve Over 24 weeks (AUC24W) | Baseline to Week 24
PK Parameter: Maximum Serum Concentration (Cmax) | Baseline up to Week 120
PK Parameter: Minimum Serum Concentration (Cmin) | Baseline up to Week 120
Time of Maximum Observed Serum Concentration (Tmax) After PDS Implant Insertion | Baseline up to Week 120
Prevalence of Anti-drug Antibodies (ADAs) at Baseline and Incidence of ADAs During the Study | Baseline up to Week 120
Prevalence of Neutralizing Antibodies at Baseline and Incidence of Neutralizing Antibodies During the Study | Baseline up to Week 120
Reported Incidence of Device Deficiencies | Baseline up to Week 120
Incidence and Severity of Ocular AEs | Baseline up to Week 120
Incidence, Severity, and Duration of AESIs | Baseline up to Week 120
Incidence, Severity, and Duration of Ocular AESIs During the Postoperative Period (up to 37 Days After Initial Implantation) and Follow-up Period (> 37 days After Implantation Surgery) | Baseline up to Week 120
Incidence and Severity of ADEs | Baseline up to Week 120
Incidence, Causality, Severity, and Duration of Anticipated Serious ADEs | Baseline up to Week 120
Substudy: Number of Participants With Ocular AESIs and Severity of Ocular AESIs After Refill-exchange Procedure | Up to approximately 72 weeks
Substudy: Duration of AESIs After Refill-exchange Procedure | Up to approximately 72 weeks
Substudy: Number of Participants With ADEs and Severity of ADEs After Refill-exchange Procedure | Up to approximately 72 weeks
Substudy: Number of Participants With Anticipated Serious ADEs After Refill-exchange Procedure | Up to approximately 72 weeks
Substudy: Duration of Serious ADEs After Refill-exchange Procedure | Up to approximately 72 weeks
Substudy: Number of Device Deficiencies After Refill-exchange Procedure | Up to approximately 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (91):
- United States (91):
  - Barnet Dulaney Perkins Eye Center, Mesa, Arizona
  - Retinal Consultants of Arizona;Opthalmology, Phoenix, Arizona
  - Arizona Retina and Vitreous Consultants, Phoenix, Arizona
  - Associated Retina Consultants, Phoenix, Arizona
  - California Retina Consultants, Bakersfield, California
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - The Retina Partners, Encino, California
  - Retina Consultants of Orange County;Clinical Research, Fullerton, California
  - Jules Stein Eye Institute/ UCLA, Los Angeles, California
  - Northern California Retina-Vitreous Associates, Mountain View, California
  - East Bay Retina Consultants, Oakland, California
  - Doheny Eye Institute, Pasadena, California
  - California Eye Specialists Medical Group, Pasadena, California
  - Retina Consultants Medical Group, Sacramento, California
  - Zuckerberg San Francisco General Hospital and Trauma Center, San Francisco, California
  - Orange County Retina Medical Group, Santa Ana, California
  - California Retina Consultants;Research Department, Santa Barbara, California
  - Eye Center of Northern Colorado, Fort Collins, Colorado
  - Colorado Clinical Research, Lakewood, Colorado
  - Retina Group of New England, Waterford, Connecticut
  - Retina Group of Florida, Fort Lauderdale, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Southern Vitreoretinal Associates;Research, Tallahassee, Florida
  - Retina Associates of Florida;Retina Associates of Florida, Tampa, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina, Marietta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Illinois Retina Associates, Joliet, Illinois
  - University Retina, Lemont, Illinois
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Retina Associates, Lenexa, Kansas
  - Retina & Vitreous Associates of Kentucky, Lexington, Kentucky
  - Maine Eye Center, Portland, Maine
  - The Retina Care Center, Baltimore, Maryland
  - Johns Hopkins Hospital;Johns Hopkins Med;Wilmer Eye Inst, Baltimore, Maryland
  - The Retina Group of Washington;Retinal Disease, Chevy Chase, Maryland
  - Cumberland Valley Retina Consultants;Clinical Research, Hagerstown, Maryland
  - Retina Specialist, Towson, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Vitreo Retinal Associates, Worcester, Massachusetts
  - Retina Specialists Of Michigan, Grand Rapids, Michigan
  - Associated Retinal Consultants - Royal Oak, Royal Oak, Michigan
  - VitreoRetinal Surgery PLLC;DBA Retina Consultants of Minnesota, Minneapolis, Minnesota
  - Pepose Vision Institute, Chesterfield, Missouri
  - Retina Institute, St Louis, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Envision Ocular, LLC, Bloomfield, New Jersey
  - Retina Associates of New Jersey, Teaneck, New Jersey
  - Long Island Vitreoretinal Consultants;Opthalmology, Great Neck, New York
  - Retina Vitreous Surgeons of Central New York, Liverpool, New York
  - New York University (NYU), New York, New York
  - Ophthalmic Consultants of Long Island, Oceanside, New York
  - Asheville Eye Associates Western Carolina Retinal Associates;Clinical Research, Asheville, North Carolina
  - Charlotte Eye Ear Nose and Throat Associates- SouthPark;Retina, Charlotte, North Carolina
  - Duke Eye Center, Durham, North Carolina
  - Graystone Eye;Clinical Research, Hickory, North Carolina
  - Cape Fear Retinal Associates, Wilmington, North Carolina
  - Cincinnati Eye Institute;Retina, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State Havener Eye Institute;Ophthalmology Research, Columbus, Ohio
  - Midwest Retina;Retina/Vitreous, Dublin, Ohio
  - Retina Vitreous Center - Glen Eagles, Edmond, Oklahoma
  - Retina Northwest;Research Department, Portland, Oregon
  - Cumberland Valley Retina Consultants, Chambersburg, Pennsylvania
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Charleston Neuroscience, Ladson, South Carolina
  - Carolina Eyecare Physicians, Mt. Pleasant, South Carolina
  - Palmetto Retina Center, West Columbia, South Carolina
  - Charles Retina Institution;Retina surgery, Germantown, Tennessee
  - Tennessee Retina, Nashville, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Texas Retina Associates, Arlington, Texas
  - Austin Research Center for Retina, Austin, Texas
  - Austin Retina Associates;Opthalmology, Austin, Texas
  - Austin Clinical Research, LLC, Austin, Texas
  - Retina & Vitreous of Texas, Bellaire, Texas
  - Texas Retina Associates;Research, Dallas, Texas
  - Texas Retina Associates, Fort Worth, Texas
  - Retina Consultants of Texas, Houston, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Rocky Mountain Retina Consultants, Murray, Utah
  - Retina Associates of Utah, PLLC;Clinical Research, Salt Lake City, Utah
  - Piedmont Eye Center, Lynchburg, Virginia
  - Wagner Kapoor Institute;Opthalmology, Norfolk, Virginia
  - Retina Institute of Virginia, Richmond, Virginia
  - Pacific Northwest Retina, Silverdale, Washington
  - Spokane Eye Clinical Research;Spokane Eye Surgery Center, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Khanani AM, Campochiaro PA, Graff JM, Marcus DM, Miller D, Mittra RA, Regillo C, Sheth VS, Bobbala A, Gune S, Lin S, Quezada-Ruiz C, Malhotra V. Continuous Ranibizumab via Port Delivery System vs Monthly Ranibizumab for Treatment of Diabetic Macular Edema: The Pagoda Randomized Clinical Trial. JAMA Ophthalmol. 2025 Apr 1;143(4):326-335. doi: 10.1001/jamaophthalmol.2025.0006. PMID 40048197
- [Derived] Stockwell AD, Chang MC, Mahajan A, Forrest W, Anegondi N, Pendergrass RK, Selvaraj S, Reeder J, Wei E, Iglesias VA, Creps NM, Macri L, Neeranjan AN, van der Brug MP, Scales SJ, McCarthy MI, Yaspan BL. Multi-ancestry GWAS analysis identifies two novel loci associated with diabetic eye disease and highlights APOL1 as a high risk locus in patients with diabetic macular edema. PLoS Genet. 2023 Aug 16;19(8):e1010609. doi: 10.1371/journal.pgen.1010609. eCollection 2023 Aug. PMID 37585454